CLINICAL TRIAL: NCT01853904
Title: Utility of Syringe Based Suction Versus Channel Suction in Bronchoalveolar Lavage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2296
Record Dates: First submitted 2013-04-05; First posted 2013-05-15 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Bronchoscopy
Keywords: Bronchoscopy; BAL; Suction
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Channel Suction first (Other): This arm is for patients who will receive channel suction first to obtain the specimen then syringe suction to obtain the specimen.
  Interventions: Procedure: Bronchoscopy/ BAL with Channel Suction; Procedure: Bronchoscopy/BAL with Syringe Suction
- Syringe Suction first (Other): This arm is for patients who will receive syringe suction first to obtain the specimen then channel suction to obtain the specimen.
  Interventions: Procedure: Bronchoscopy/ BAL with Channel Suction; Procedure: Bronchoscopy/BAL with Syringe Suction

INTERVENTIONS:
Procedure: Bronchoscopy/ BAL with Channel Suction — The wall suction used for the channel suction will be set at 80 mm Hg. This arm is for patients who will receive channel suction first to obtain the specimen then syringe suction to obtain the specimen.
Procedure: Bronchoscopy/BAL with Syringe Suction — Syringe based suctioning will be performed with 20mL syringe.

SUMMARY:
Bronchoalveolar lavage (BAL) is a common technique among pulmonologists. Its goal is to collect cells from alveolar units. This is done by wedging a flexible bronchoscope in a bronchus, instilling saline, and removing the saline via suction. Two techniques are currently used for suctioning: syringe based and channel suction.

The investigators concern is that channel suction creates too much force and there is collapsing of the airways which results in decreased fluid removal as well as cell sampling. The investigators propose that syringe based suctioning will not only return more of the instilled fluid but also more cells from the alveoli.

DETAILED DESCRIPTION:
The pulmonary segment with the most disease on imaging will be the segment sampled. The scope will be wedged in the airway leading to that segment and 100mL of saline will be instilled into the selected segment and collected via the syringe based or channel based suction. Prior to unwedging, another 100mL of saline will be instilled into the same segment and will be collected using the alternative method. There will not be randomization, but the investigators will alternate which method is used first to eliminate confounding variables. All patients will receive both modalities of suctioning. The wall suction used for the channel suction will be set at 80 mm Hg. Syringe based suctioning will be performed with 20mL syringe. Total amount of fluid collected will be recorded and samples will be sent for cell count and differential as well as Gram stain and culture. Results of the two techniques will then be compared to determine which is the superior suctioning modality for BAL.

ELIGIBILITY:
Inclusion Criteria:

* Bronchoscopy scheduled

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of Syringe Suction versus Channel Suction to retrieve volume | 24 hours

SECONDARY OUTCOMES:
Efficacy of Syringe suction versus Channel suction to retrieve alveolar cells | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Brent Brown, MD, Principal Investigator — OUHSC
Locations (1):
- OUHSC, Oklahoma City, Oklahoma, United States